CLINICAL TRIAL: NCT03547765
Title: Assessment of Sexual Health of Obese Men Before and After Paresis Bariatric Surgery. Prospective Multicentre Study.
Brief Title: Sexual Health of Obese Men Before and After Bariatric Surgery.
Acronym: BARIASSO
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/06
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Bariatric Surgery
Keywords: Obesity; Sexual Dysfunction
MeSH Terms: conditions — Obesity; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Compare Male Health Sexual Questionnaire (MHSQ) before and after bariatric surgery to assess the sexual health of the obese men with a recommended and exhaustive tool. There are few data that evaluate the sexual health of this population.

DETAILED DESCRIPTION:
The sexual dysfunctions are more commonly in the obese men population. For example, erectile dysfunction is more than twice as common as in the general population. However, the data on sexuality in the broad sense are rarer. The latter are in favor of an inconsistent improvement and use the Brief Male Sexual Function Inventory. The MHSQ is now recommended by the French Urology Association to evaluate more fully male sexuality. Its relatively recent validation explains the few studies referring to. The investigators believe that one of the major determinants of sexual health in obese men is the self-image.

The investigators will submit to the patients the male heath sexual questionnaire, the Beck Depression Inventory (BDI) and the Multidimensional Body Self Relations Questionnaire - Appearance Scales (MBSRQ-AS) and collect weight, BMI and age during the classic follow up. The data will be collected during the preoperative assessment as well as 6 months and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Any male patient eligible for bariatric surgery, the indication of which was decided at a multidisciplinary consultation meeting.
* not opposed to research.
* benefiting from social security cover.

Exclusion Criteria:

- inclusion criteria not satisfied

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The sexual dysfunctions are more commonly in the obese men population. For example, erectile dysfunction is more than twice as common as in the general population.
Study Population: The sexual dysfunctions are more commonly in the obese men population. There are few data that evaluate the sexual health of this population. We believe that one of the major determinants of sexual health in obese men is the self-image.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Average of Male Health Sexual Questionnaire (MHSQ) score | At 12 month after inclusion day
  Comparison of MHSQ score before and after bariatric surgery to assess the sexual health of the obese men. MHSQ measures differents aspects of ability to have sexual activities: erection, ejaculation and satisfaction.
  MHSQ score varies from 0, extremely embarrassed, to 90, not at all embarrassed.

SECONDARY OUTCOMES:
Correlation between Male Health Sexual Questionnaire (MHSQ) score and Multidimensional Body Self Relations Questionnaire - Appearance Scales (MBSRQ-AS) score | At 12 month after inclusion day
  Correlation investigation between MHSQ score and MBSRQ-AS score
Correlation between Beck Depression Inventory (BDI) score and Multidimensional Body Self Relations Questionnaire - Appearance Scales (MBSRQ-AS) score | At 12 month after inclusion day
  Correlation investigation between MBSRQ-AS score and BDI score
Correlation between Beck Depression Inventory (BDI) score and Male Health Sexual Questionnaire (MHSQ) score | At 12 month after inclusion day
  Correlation investigation between BDI score and MHSQ score

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Mutualiste de Pessac, Pessac
  - Hôpital Haut-Lévêque - groupe hospitalier Sud, Pessac